CLINICAL TRIAL: NCT01252914
Title: A Prospective Evaluation of Open-angle Glaucoma Subjects on Two Topical Hypotensive Medication Treated With One Suprachoroidal Stent
Brief Title: A Prospective Evaluation of Open-Angle Glaucoma Subjects on Two Topical Hypotensive Medications Treated With One Suprachoroidal Stent
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCF-019
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Subject With Primary Open-angle Glaucoma (POAG)
Keywords: Open angle; Glaucoma; Surgery; Ocular Hypertension; Eye Diseases
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Eye Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- One iStent Supra Stent and medication (Experimental): The study assesses the efficacy and safety of one iStent Supra stent in the reduction of intraocular pressure associated with primary open-angle glaucoma
  Interventions: Device: iStent Supra Stent

INTERVENTIONS:
Device: iStent Supra Stent — Implantation of one iStent Supra Stent through a small temporal clear corneal incision

SUMMARY:
The purpose of this study is to assess the efficacy and safety of one iStent supra stent in the reduction of intraocular pressure associated with primary open-angle glaucoma.

DETAILED DESCRIPTION:
The study assesses the efficacy and safety of one iStent supra stent in the reduction of intraocular pressure associated with primary open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary open-angle glaucoma (POAG)
* Subjects on two topical hypotensive medications

Exclusion Criteria:

* Traumatic, uveitic, neovascular, or angle closure glaucoma
* Fellow eye already enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-12 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Mean diurnal Intraocular Pressure reduction of greater than or equal to 20% at month 12 vs. baseline | 12 months

SECONDARY OUTCOMES:
Mean diurnal Intraocular Pressure < 18 mmHg at month 12 | 12 months

OTHER OUTCOMES:
Safety | 0-61 months
  Rate of ocular adverse events through 61 months
  * Findings from Intraocular Pressure, best corrected visual acuity, visual field, specular microscopy measurements
  * Findings from slit-lamp, fundus and gonioscopic examinations

CONTACTS AND LOCATIONS:
Overall Officials: Lilit Voskanyan, MD, Principal Investigator — SV Malayan Ophthalmological Center, Yerevan, Armenia
Locations (1):
- S.V. Malayan Ophthalmology Centre, Yerevan, Armenia